CLINICAL TRIAL: NCT05713032
Title: High-voltage Fluoroscopic Guided Pulsed Radiofrequency in Comparison With Standard-voltage Pulsed Radiofrequency on Dorsal Root Ganglion in Chronic Lumbosacral Radicular Pain
Brief Title: Pulsed Radiofrequency in Chronic Lumbosacral Radicular Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mina Nabil Habib, doctor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E/C. S/N. T124/2022
Record Dates: First submitted 2023-01-24; First posted 2023-02-06 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Lumbar Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard voltage group (Active Comparator): The Standard voltage group will be given a onetime pulsed radiofrequency (PRF) therapy. All subjects in this group will be given radiofrequency therapy on the dorsal root ganglion using the same tools and procedures by the same operator. Pulsed RF mode of RF generator will be used with following parameters --Temperature 42°C -- Frequency 2 Hertz - Pulse Width 20msec-Amplitude output voltage 45 Volt for Duration of 480sec done in 2 cycles.
  Interventions: Procedure: Pulsed radiofrequency on lumbar dorsal root ganglion
- high voltage group (Active Comparator): The High voltage group will be given a onetime pulsed radiofrequency (PRF) therapy. All subjects in this group will be given radiofrequency therapy on the dorsal root ganglion using the same tools and procedures by the same operator. Pulsed RF mode of RF generator will be used with following parameters --Temperature 42°C -- Frequency 2 Hertz - Pulse Width 20msec-Amplitude output voltage will be gradually increased to reach the highest voltage for each patient (55-75 Volt) for Duration of 480sec done in 2 cycles.
  Interventions: Procedure: Pulsed radiofrequency on lumbar dorsal root ganglion

INTERVENTIONS:
Procedure: Pulsed radiofrequency on lumbar dorsal root ganglion — voltage of pulsed radiofrequency on DRG

SUMMARY:
To evaluate the efficacy of usage of High-voltage pulsed radiofrequency on DRG in comparison to standard-voltage pulsed radiofrequency intervention in patients with chronic lumbosacral radicular pain

DETAILED DESCRIPTION:
Lumbosacral radicular (LRS) pain is one of the most common health care problem. Up to 5% of the population older than 30 years of age suffer low back pain radiating into the leg, making it probably the most commonly occurring form of neuropathic pain.

Radicular pain has been discerned as the pain arising in a limb or trunk which is caused by ectopic activation of nociceptive afferent fibers in a spinal nerve or its roots or other neuropathic mechanisms. More accurately, radicular pain is a term applied to describe pain that results from the stimulation of, or a disorder of, a nerve root.

Acute lumbosacral radicular pain, caused by disc herniation, improves considerably in the short-term. About three quarters of patients will have symptoms of recovery within 3 months; however, there is a high recurrence rate, and when pain persists after this period the prognosis is rather unfavorable, especially in the female population. Conservative therapy (pharmacotherapy or physiotherapy) is effective in 60% of cases, while the rest of cases progress into chronic pain. This results in a high degree of disability and ending with higher medical expenses.

Patients suffering lumbosacral radicular pain often experience a reduced functionality leading to incapacity to work. A quarter of patients are still out of work 2 years after onset.

Despite its high prevalence and significant impact on quality of life, the optimal conservative treatment for patients with radicular pain is not known. Considering the moderate quality of published evidence, the efficacy and tolerability of pharmacological treatment in primary care for patients with lumbosacral radicular pain is unclear.

In the DRG, there is a process that takes place after being compressed by disc prolapse where a cascade of events within the DRG and upstream within the dorsal horn (DH) of the spinal cord leads to constitutive release of cytokines, production of abnormal ion channels, abnormal ion currents, early and late gene changes, and the development of chronic neuropathic pain. With this knowledge regarding the role of DRG neurons and non-neuronal cells within the DRG in the genesis of neuropathic pain, pharmacologic agents such as tetrodotoxin and non-pharmacologic treatments for neuropathic pain including electrical stimulation (neuromodulation) therapies targeting the DRG have been or are being developed.

Pulsed radiofrequency (PRF) is a therapeutic strategy that has been used by pain practitioners as a non- or minimally autodestructive technique in which short bursts of high-frequency current are applied to nervous tissue.

PRF is delivered in a pulse of 20 ms followed by a silent period of 480 ms to avoid radiofrequency heat lesions, and Pulsed radiofrequency (PRF) treatment uses high-frequency current intermittently and its use adjacent to the dorsal root ganglion (DRG) has been suggested for the treatment of radicular pain.

It was previously demonstrated in other studies that the therapeutic effectiveness of PRF is affected by its parameters and the high-voltage PRF has been promising to enhance the clinical therapeutic effectiveness significantly for patients with neuralgia

ELIGIBILITY:
Inclusion Criteria:

1. More than 18 years old
2. Radiating Leg pain (with or without low back pain)
3. Unresponsiveness or partial response to oral medications, physical therapy
4. Confirmed by clinical examination and lasting for > 6 months with preoperative Numeric Rating Scales (NRS) score more than 4
5. Clinical presentation confirmed by Magnetic resonance imaging showing neural compression.

Exclusion Criteria:

1. Blood coagulopathies
2. Infection at the site of puncture,
3. History of mental disorder
4. History of drug abuse
5. MRI not consistent with clinical symptoms
6. Radiculopathies with significant motor deficits requiring urgent surgery (e.g., Cauda Equina syndrome).
7. Patients affected by central neurological impairment or peripheral distal neuropathies in the lower limbs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale | 6 months
  Numeric scale used to evaluate pain severity with 0 as the lowest score (no pain at all) and 10 as the highest score (most serious pain beyond endurance)

SECONDARY OUTCOMES:
Oswestry low back disability questionnaire | 6 months
  Questionnaire composed of ten questions and for each question, there is a possible points; 0 for the first answer, 1 for the second answer, etc.
  Score 0-4 : No disability Score 5-14 : Mild disability Score 15-24 : Moderate disability Score 25-34 : Severe disability Score 35-50 : Completely disabled

OTHER OUTCOMES:
Record of Complications intra or post-intervention | 6 months
  as infection (eg; Epidural abscess , diskitis ) , bleeding , dural puncture and nerve injury

CONTACTS AND LOCATIONS:
Overall Officials: Sahar A Elkaradawy, professor, Study Director — yes; Mohamed H Ellakany, professor, Study Director — yes
Locations (1):
- Medical Research Institute, Alexandria, Al, Egypt

REFERENCES:
- [Result] Cohen SP, Greuber E, Vought K, Lissin D. Safety of Epidural Steroid Injections for Lumbosacral Radicular Pain: Unmet Medical Need. Clin J Pain. 2021 Sep 1;37(9):707-717. doi: 10.1097/AJP.0000000000000963. PMID 34265792
- [Result] Krames ES. The role of the dorsal root ganglion in the development of neuropathic pain. Pain Med. 2014 Oct;15(10):1669-85. doi: 10.1111/pme.12413. Epub 2014 Mar 18. PMID 24641192
- [Result] Kim SJ, Park SJ, Yoon DM, Yoon KB, Kim SH. Predictors of the analgesic efficacy of pulsed radiofrequency treatment in patients with chronic lumbosacral radicular pain: a retrospective observational study. J Pain Res. 2018 Jun 26;11:1223-1230. doi: 10.2147/JPR.S164414. eCollection 2018. PMID 29983585
- [Result] Lee DG, Cho YW, Ahn SH, Chang MC. The Effect of Bipolar Pulsed Radiofrequency Treatment on Chronic Lumbosacral Radicular Pain Refractory to Monopolar Pulsed Radiofrequency Treatment. Pain Physician. 2018 Mar;21(2):E97-E103. PMID 29565952
- [Result] Marliana A, Yudianta S, Subagya DW, Setyopranoto I, Setyaningsih I, Tursina Srie C, Setyawan R, Rhatomy S. The efficacy of pulsed radiofrequency intervention of the lumbar dorsal root ganglion in patients with chronic lumbar radicular pain. Med J Malaysia. 2020 Mar;75(2):124-129. PMID 32281592
- [Result] Van Boxem K, van Bilsen J, de Meij N, Herrler A, Kessels F, Van Zundert J, van Kleef M. Pulsed radiofrequency treatment adjacent to the lumbar dorsal root ganglion for the management of lumbosacral radicular syndrome: a clinical audit. Pain Med. 2011 Sep;12(9):1322-30. doi: 10.1111/j.1526-4637.2011.01202.x. Epub 2011 Aug 3. PMID 21812907
- [Result] Vanneste T, Van Lantschoot A, Van Boxem K, Van Zundert J. Pulsed radiofrequency in chronic pain. Curr Opin Anaesthesiol. 2017 Oct;30(5):577-582. doi: 10.1097/ACO.0000000000000502. PMID 28700369
- [Result] Vigneri S, Sindaco G, La Grua M, Zanella M, Lo Bianco G, Paci V, Vinci FM, Sciacca C, Ravaioli L, Pari G. Electrocatheter-mediated High-voltage Pulsed Radiofrequency of the Dorsal Root Ganglion in the Treatment of Chronic Lumbosacral Neuropathic Pain: A Randomized Controlled Study. Clin J Pain. 2020 Jan;36(1):25-33. doi: 10.1097/AJP.0000000000000766. PMID 31577546
- [Result] Wan C, Dong DS, Song T. High-Voltage, Long-Duration Pulsed Radiofrequency on Gasserian Ganglion Improves Acute/Subacute Zoster-Related Trigeminal Neuralgia: A Randomized, Double-Blinded, Controlled Trial. Pain Physician. 2019 Jul;22(4):361-368. PMID 31337167
- [Result] Wan CF, Liu Y, Dong DS, Zhao L, Xi Q, Yu X, Cui WY, Wang QS, Song T. Bipolar High-Voltage, Long-Duration Pulsed Radiofrequency Improves Pain Relief in Postherpetic Neuralgia. Pain Physician. 2016 Jul;19(5):E721-8. PMID 27389115
- [Result] Yang S, Kim W, Kong HH, Do KH, Choi KH. Epidural steroid injection versus conservative treatment for patients with lumbosacral radicular pain: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2020 Jul 24;99(30):e21283. doi: 10.1097/MD.0000000000021283. PMID 32791709